CLINICAL TRIAL: NCT04202705
Title: A First-in-human Dose-escalation and Expansion Study With the Antibody-drug Conjugate SYD1875 to Evaluate the Safety, Pharmacokinetics and Efficacy in Patients With 5T4-expressing Locally Advanced or Metastatic Solid Tumours
Brief Title: A First-in-human Dose-escalation and Expansion Study With the Antibody-drug Conjugate SYD1875
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Byondis B.V. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: SYD1875.001
Record Dates: First submitted 2019-12-12; First posted 2019-12-17 (Actual); Last update posted 2023-01-30 (Actual); Status verified 2023-01

CONDITIONS: Solid Tumor
Keywords: ADC; 5T4; solid tumors; duocarmycin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SYD1875 (Experimental): 5T4-targeting Antibody-Drug Conjugate
  Interventions: Drug: SYD1875

INTERVENTIONS:
Drug: SYD1875 — SYD1875 IV (in the vein) infusion every three weeks. Number of cycles: until cancer progression or unacceptable toxicity develops. Different doses.

SUMMARY:
This is the first-in-human study with SYD1875, an antibody-drug conjugate (ADC) comprising of a humanized IgG1 monoclonal antibody directed against the 5T4 oncofetal antigen covalently conjugated to a duocarmycin-based linker-drug. This study includes a dose-escalation part (Part 1) in which the maximum tolerated dose (MTD) and recommended dose for expansion (RDE) will be determined, and an expansion part (Part 2) to evaluate efficacy and safety in specific patient cohorts.

DETAILED DESCRIPTION:
Cancer cells can have different kinds of proteins on their cell surface; one of these is the oncofetal antigen 5T4. 5T4 plays an important role in the development of cancer. Currently no drugs are available that work via the 5T4 antigen.

The new cancer drug SYD1875 is being developed by Byondis B.V. SYD1875 is an antibody-drug conjugate and consists of two parts: an antibody and a linker-drug moiety containing a toxin. The antibody part binds to 5T4 on the surface of the cancer cell. When SYD1875 binds to this cancer cell, it will be internalized by the cell. After proteolytic cleavage of the linker, the toxin will be split off in the cell and the cancer cell will be killed. Thus, SYD1875 can be considered as a form of targeted chemotherapy.

This is the first study in which SYD1875 is administered to humans. The study consists of two parts:

Part 1 is the dose-escalation part in which a low dose of SYD1875 is given to cancer patients. If it is well tolerated, a higher dose of SYD1875 will be given to other cancer patients until the maximum tolerated dose is reached.

In Part 2 of the study, groups of patients with a specific type of cancer will receive the SYD1875 dose which has been selected for further evaluation.

All patients from both parts of the study will receive SYD1875 infusions every three weeks until progression of the cancer or unacceptable toxicity develops.

ELIGIBILITY:
Main Inclusion Criteria:

* Patient with histologically-confirmed, locally advanced or metastatic cancer who has progressed on standard therapy or for whom no standard therapy exists, with the following restriction:
* Part 1: solid tumours of any origin
* Part 2: three patient cohorts
* Tumour 5T4 membrane staining according protocol
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 1;
* Adequate organ function
* For Part 2: measurable disease

Main Exclusion Criteria:

* Having been treated with:

  1. 5T4-targeting therapy at any time
  2. Trastuzumab duocarmazine (SYD985) at any time
  3. Other anticancer therapy within 4 weeks or as defined in the protocol
  4. Hormone therapy within 1 week
* History or presence of keratitis, clinically significant renal disease, lung disease, or cardiovascular disease as specified in the protocol
* Symptomatic brain metastases, brain metastases requiring steroids or treatment for brain metastases within 8 weeks

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 31 (Actual)
Dates: Start 2020-02-28 (Actual); Primary Completion 2022-06-22 (Actual); Study Completion 2023-01-26 (Actual)

PRIMARY OUTCOMES:
Incidence of dose-limiting toxicities | 21 days
  Part 1

SECONDARY OUTCOMES:
Objective response rate | 21 days
  Part 2

CONTACTS AND LOCATIONS:
Overall Officials: Ellen Mommers, PhD, Study Director — Byondis B.V., The Netherlands
Locations (3):
- Institut Jules Bordet, Brussels, Belgium
- France (2):
  - Institut Bergonié, Bordeaux
  - Centre Oscar Lambret, Lille

IPD SHARING:
Plan to Share IPD: No